CLINICAL TRIAL: NCT00002027
Title: Protocol For the Treatment of Cryptosporidiosis in AIDS Patients With Diclazuril (R64,433)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Janssen, LP (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 038A; JRD 64,433/1101
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-06

CONDITIONS: Cryptosporidiosis; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Cryptosporidiosis; Diarrhea; diclazuril; Coccidiostats; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Cryptosporidiosis; HIV Infections; AIDS-Related Opportunistic Infections; Diarrhea; Acquired Immunodeficiency Syndrome | interventions — diclazuril

INTERVENTIONS:
Drug: Diclazuril

SUMMARY:
To evaluate the safety and efficacy of diclazuril capsules compared with placebo capsules as treatment of cryptosporidial related diarrhea in AIDS patients. Treatment efficacy will be based on the drug's clinical results and on its anti-protozoan effects. Safety will be assessed by the occurrence of side effects as reported by patients at their visits and by frequent monitoring of hematology, biochemistries, and urinalysis.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Patients who require anti-diarrheal medication must have received only one anti-diarrheal medication, loperamide, for at least 7 days prior to study entry. Dose of loperamide cannot be increased during study.
* Aerosolized pentamidine.
* Ganciclovir for cytomegalovirus (CMV) retinitis only but patient must be stable at least 4 weeks prior to study entry.
* Zidovudine (AZT).
* Nystatin for oropharyngeal infections if not taken within 2 hours of diclazuril.

Patients must have:

* Diagnosis of AIDS that is confirmed HIV positive by Western blot or AIDS defined diagnosis, or CDC defined AIDS. Stool specimens positive for cryptosporidium oocysts.
* Given written informed consent after the purpose and nature of the study, as well the possible drug-related adverse effects, have been explained.
* Ability to return for all subsequent applicable visits on days 8, 15, 21, and, if necessary, 28.

Prior Medication:

Allowed:

* Aerosolized pentamidine.
* Loperamide.
* Ganciclovir for cytomegalovirus (CMV) retinitis.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Diagnosis of cryptosporidiosis less than 4 weeks prior to study entry, unless patient has been diagnosed with AIDS for more than 4 weeks.
* Other treatable enteric pathogens including Clostridia must be treated and eradicated prior to study entry.
* Inability to swallow capsules.
* Uncontrolled vomiting.

Concurrent Medication:

Excluded:

* Trimethoprim/sulfamethoxazole (Bactrim).
* Ganciclovir for any other reason except cytomegalovirus (CMV) retinitis.
* Other antibiotics.
* Other anti-protozoal drugs.
* Anti-fungal drugs other than nystatin.
* Amphotericin B.
* Other investigational drugs.

Patients with the following are excluded:

* Diagnosis of cryptosporidiosis less than 4 weeks prior to study entry, unless patient has been diagnosed with AIDS for more than 4 weeks.
* Inability to swallow capsules.
* Uncontrolled vomiting.
* Life expectancy of < 28 days.
* Can not be depended upon to follow the instructions of the investigator.
* Participation in an investigational study within 15 days of study entry.

Prior Medication:

Excluded within 15 days of study entry:

* Another investigational drug or device (except aerosolized pentamidine).

Prior Treatment:

Excluded within 15 days of study entry:

* Participation in an investigational study.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Dr Douglas Dieterich, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York

REFERENCES:
- [Background] Connolly GM, Youle M, Gazzard BG. Diclazuril in the treatment of severe cryptosporidial diarrhoea in AIDS patients. AIDS. 1990 Jul;4(7):700-1. doi: 10.1097/00002030-199007000-00020. No abstract available. PMID 2397069
- [Background] Soave R, Dieterich D, Kotler D, Gassyuk E, Tierney AR, Liebes L, Legendre R. Oral diclazuril therapy for cryptosporidiosis. Int Conf AIDS. 1990 Jun 20-23;6(1):252 (abstract no ThB520)